CLINICAL TRIAL: NCT03212586
Title: Randomized, Placebo-controlled, Double-blind, Parallel-group Study to Investigate the Safety, Tolerability and Pharmacokinetics of Increasing Single Oral Doses of BAY1902607 Including the Relative Bioavailability Between Different Pharmaceutical Formulations and the Effect of Food on the Pharmacokinetics of BAY1902607 in Healthy Men
Brief Title: BAY 1902607: Single Dose Escalation, Safety and Tolerability, Pharmacokinetics, Bioavailability, Food Effect
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 18922; 2017-000978-11 (EudraCT Number)
Record Dates: First submitted 2017-07-07; First posted 2017-07-11 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Clinical Trials, Phase I as Topic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dose escalation BAY1902607 (Experimental): Dose 1 to 9 of BAY1902607
  Interventions: Drug: BAY1902607
- Dose escalation Placebo (Placebo Comparator): Dose 1 to 9 of matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BAY1902607 — Escalating doses of BAY1902607; single dose administration; different dosage forms (redosing of BAY1902607 at dose group 4 with different formulations; redosing of BAY1902607 solid formulation at dose group 4 together with food)
  Arms: Dose escalation BAY1902607
Drug: Placebo — Escalating doses of Placebo; single dose administration; different dosage forms (redosing of Placebo at dose group 4 with different formulations; redosing of Placebo solid formulation at dose group 4 together with food)
  Arms: Dose escalation Placebo

SUMMARY:
This study is a first-in-man study that will investigate the safety, tolerability and pharmacokinetics of ascending single doses of BAY1902607 using a placebo controlled, randomized, single center design. In addition the influence of food on the pharmacokinetics of BAY1902607 and the bioavailability between different pharmaceutical formulations will be investigated

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects.
* Age: 18 to 45 years (inclusive) .
* Body mass index (BMI) : ≥18 and ≤30 kg/m^2.
* Race: White.

Exclusion Criteria:

* Any findings from the medical examination (including medical history, physical examination, vital signs, laboratory tests and ECG) deviating from normal and deemed by the investigator to be of clinical relevance.
* Relevant diseases within the 4 weeks before the first drug administration.
* Febrile illness within the week before the first taste test is conducted.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2017-07-18 (Actual); Primary Completion 2018-05-03 (Actual); Study Completion 2018-07-27 (Actual)

PRIMARY OUTCOMES:
Number of subjects with treatment-emergent adverse events | Up to 11 weeks
  AE is any untoward medical occurrence (i.e. any unfavorable and unintended sign [including abnormal laboratory findings], symptom or disease) in a patient or clinical investigation subject after providing written informed consent for participation in the study. AEs (except for those in the 60 mg dose group) were considered to be treatment-emergent if they had started or worsened within the interval from first study drug administration until the follow-up visit. For the 60 mg dose group, AEs were considered to be TEAEs if they had started or worsened within one of the following intervals: 1) from first administration of study medication in treatment period 1 to 15 days thereafter, 2) from second administration of study medication in treatment period 2 to 15 days thereafter, 3) from third administration of study medication in treatment period 3 to follow-up visit.
Number of subjects with severity of treatment-emergent adverse events | Up to 11 weeks
  AEs were considered to be TEAEs if they had started or worsened within the interval from first study drug administration until the follow-up visit (except for the 60 mg dose group: from first study drug administration in treatment period 1 to 15 days thereafter; from second study drug administration in treatment period 2 to 15 days thereafter; from third study drug administration in treatment period 3 to follow-up visit). Classification of the intensity: Mild (usually transient and might have required only minimal treatment or therapeutic intervention, did not generally interfere with usual activities of daily living), Moderate (usually alleviated with additional specific therapeutic intervention, interfered with usual activities of daily living, causing discomfort but posed no significant or permanent risk of harm to the research subject), Severe (required intensive therapeutic intervention, interrupted usual activities of daily living, or significantly affected clinical status).

CONTACTS AND LOCATIONS:
Locations (1):
- CRS Clinical Research Services Berlin GmbH, Berlin, Germany

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe. — http://www.clinicaltrialsregister.eu/